CLINICAL TRIAL: NCT01118676
Title: Phase I Trial Evaluating Continuous Infusion of Cilengitide Together With Radiochemotherapy in Patients With Locally Advanced Non Small Cell Lung Cancer
Brief Title: Cilengitide Together With Radiochemotherapy in Patients With Locally Advanced Non Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07 POUM 01
Record Dates: First submitted 2010-05-05; First posted 2010-05-07 (Estimated); Last update posted 2022-05-24 (Actual); Status verified 2015-09

CONDITIONS: Locally Advanced Non Small Cell Lung Cancer (NSCLC)
Keywords: locally advanced non small cell lung cancer (NSCLC), locally advanced, Phase I, Cilengitide, concomitant radiochemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cilengitide; Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cilengitide with standard radiochemotherapy (Experimental): Cilengitide (4 dose levels are defined :12, 18, 27 et 40 mg /hour) concomitant with radiotherapy (standard radiotherapy of 66 Gy, 2 Gy per daily fraction) and cisplatin and vinorelbine based chemotherapy.
  Interventions: Drug: cilengitide, radiochemotherapy

INTERVENTIONS:
Drug: cilengitide, radiochemotherapy — Cilengitide will be administered alone as continuous infusion two weeks before the radiochemotherapy and will then be continued during radiochemotherapy (standard radiotherapy of 66 Gy, 2 Gy per daily fraction, and cisplatin and vinorelbine based chemotherapy)as continuous infusion.
  The dose levels investigated will be applied to the continuous administration of cilengitide(a maximum of 4 dose levels : 12, 18, 27 et 40 mg /hour).
  After the end of concomitant radiochemotherapy, cilengitide will be administered i.v. at a dose of 2000 mg twice weekly until the end of chemotherapy.

SUMMARY:
This is a two-center study which includes 24 patients maximum on 36 months : 24 months accrual - 12 months follow up.

Eligible patients are included according to a standard 3+3 design.

Patients included in the trial will be treated with a combination of radiochemotherapy (standard radiotherapy of 66 Gy, 2 Gy per daily fraction, and cisplatin and vinorelbine based chemotherapy).

Cilengitide will be administered alone as continuous infusion two weeks before the radiochemotherapy and will then be continued during radiochemotherapy as continuous infusion.

The dose levels investigated will be applied to the continuous administration (a maximum of 4 dose levels).

After the end of concomitant radiochemotherapy, cilengitide will be administered i.v. at a dose of 2000 mg twice weekly until the end of chemotherapy.

The dose of Cilengitide administered after radiotherapy will not be increased. 4 dose levels are defined:12, 18, 27 et 40 mg /hour.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven non small cell lung cancer
2. Inoperable tage IIIA or IIIB non small cell lung cancer
3. Age ≥ 18 years
4. PerfLife expectancy ≥6 months
5. Hematological function : neutrophils ≥1500/mm3 and platelets ≥ 100000/mm3
6. Hepatic function: Bilirubin within normal limits et AST and ALT ≤ 2 times the upper limit of normal (ULN).
7. Renal function: Creatinine ≤ 1.5 times ULN.
8. Absence of cardiac insufficiency, absence of unstable angina, absence of arrythmia
9. Patient has health insurance coverage.
10. Signed informed consent.

Exclusion Criteria:

1. Patients previously treated for a malignancy by means of chemotherapy, radiotherapy or surgery.
2. Uncontrolled hypertension
3. Uncontrolled bleeding within the last 3 months.
4. Patients under anti-coagulation with anti-vitamin K or therapeutic dose heparin ; low-molecular heparins for prophylaxis are permitted and are not considered an exclusion criterion.
5. Presence of cerebral metastases.
6. Participation in a clinical trial within the last 8 weeks.
7. Any other specific concomitant anti-tumor treatment (such as chemotherapy, radiotherapy …).
8. Patients with a history of myocardial infarction or a cerebral vascular accident within the last 12 months.
9. Continued use of aspirin (>325mg/day)
10. Major surgery whiting the last 28 days or planned.
11. Major non-healing wound, ulcer
12. Pregnant or breastfeeding women cannot participate in this trial. Women of reproductive potential must have a negative pregnancy test (blood) within 72 hours before the start of treatment.
13. Men and women of reproductive potential must use an efficient contraceptive method when entering the trial and until one months after the end of treatment.
14. History of a thrombo-embolic or hemorrhagic event.
15. Patients put under tutelage.
16. Patients not able to follow the procedures visits, exams foreseen by the trial.
17. Any other severe medical or psychiatric condition or biological anomaly - acute or chronic - that, in the investigator's opinion - may render the inclusion of the patient inappropriate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
To determine the Maximum Tolerated dose (MTD) of Cilengitide administered as continuous infusion during standard radiochemotherapy | at the end of the trial

SECONDARY OUTCOMES:
To determine the rate of objective response according to RECIST and pathological response. | at the end of the trial
To determine the survival free of metastases and the survival without local relapse at one year. | at the end of the trial
To determine the overall survival | at the end of the trial
To determine the toxicity of the combination of radiochemotherapy and continuous infusion cilengitide as well as the toxicity of the combination of chemotherapy and twice weekly cilengitide. | at the end of the trial
Ancillary studies will be undertaken to determine factors predictive of response to treatment and to characterize the anti-angiogenic effect of Cilengitide. | at the end of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth COHEN-JONATHAN MOYAL, Pr, Principal Investigator — Institut Claudius Regaud
Locations (2):
- France (2):
  - CHU Toulouse Larrey, Toulouse
  - Institut Claudius Regaud, Toulouse